CLINICAL TRIAL: NCT04652635
Title: Management of Nailbed Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Luan, Resident in Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59042
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Nail Bed Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: 6 month appearance will be assessed by a blinded individual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nail plate removal, nail bed repair (Active Comparator): Participants will undergo nail plate removal and nail bed repair, and follow up at clinic visits at 1 week, 3 months, and 6 months
  Interventions: Procedure: Nail plate removal, nail bed repair
- Observation (No Intervention): Participants will follow up at clinic visits at 1 week, 3 months, and 6 months

INTERVENTIONS:
Procedure: Nail plate removal, nail bed repair — Injection of local anesthetic, removal of nail plate, inspection of nail bed, repair of nail bed with suture and/or adhesive
  Arms: Nail plate removal, nail bed repair

SUMMARY:
The purpose of the study is to determine whether nail plate removal in suspected nailbed injury improves patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* any individual greater than or equal to 2 years of age presenting with a suspected nailbed injury (laceration adjacent to or through nail plate and/or subungual hematoma) with the nail plate present

Exclusion Criteria:

* nail plate absent over the nailbed injury

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience complications over time | 6 months
  Any complication, including but not limited to infection or wound healing complications
Change in pain score over time as measured on a pain scale | 6 months
  Scored from 0-10 (higher scores indicate worse pain)
Change in cosmetic appearance over time as measured by the Oxford Finger Nail Appearance Score | 6 months
  Oxford Finger Nail Appearance Score (OFNAS), ranges from 0 to 5 (5 is the best appearance)
Change in upper extremity function over time as measured by the QuickDash score | 6 months
  Quick Disabilities of Arm, Shoulder, & Hand (QuickDASH) score, ranges from 0 (no disability) to 100 (most severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Luan, MD, Principal Investigator — Stanford University; Jeffrey Yao, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No